#### Fred Hutchinson Cancer Research Center

## Consent to take part in a research study:

## The Air Study

Principal Investigator: Trang VoPham, PhD, MS. Fred Hutchinson Cancer Research

Center. 206-667-2642

## Important things to know about this study.

You are invited to participate in a research study. The purpose of this research is to provide people with information regarding their air pollution exposure, its health effects, and strategies to reduce personal exposure to air pollution.

People who agree to join the study will be asked to complete 2 online questionnaires, watch 2 educational videos about air pollution, its health effects, and exposure mitigation strategies, and use a wearable air pollution sensor over the course of 5 weeks.

You do not have to join this study. Although the study will not benefit participants directly, we hope to use the information that we gather to develop larger studies to help people increase their knowledge and awareness of the harmful health effects of air pollution. The study procedures are associated with a very small risk for compromised confidentiality inherent in data collection, as described below in this form.

The Prevent Cancer Foundation® is paying for this research to be done.

The following is a more complete description of this study. Please read this description carefully. You can ask any questions you want to help you decide whether to join the study. If you join this study, we will give you a signed copy of this form to keep for future reference

## We would like you to join this research study.

We are conducting a research study to determine if providing people with information regarding their air pollution exposure using wearable sensors, the harmful health effects of air pollution, and exposure mitigation strategies will increase knowledge of air pollution and promote preventive health behaviors to reduce personal air pollution exposure.

Since you are a healthy adult (age 18-64 years) living in the Seattle metropolitan area, own a smartphone, are not traveling outside of King County for more than 2 consecutive days in the next 2 months, and leave your home for at least 7 hours per week, we would

FHCRC IRB Approval AUG 13 2021 Document Released Date like to ask you to join this study. We will enroll up to 20 people. Although the study will not benefit participants directly, we hope the information we learn will help people increase knowledge and awareness of their personal air pollution exposure.

If you agree to be in this study, you will do the following:

**Questionnaires**: You will complete 2 online questionnaires asking about demographics, health and lifestyle factors, locations, knowledge about air pollution and health effects, and air pollution preventive health behaviors. There is one questionnaire to be completed during week 1 of the study, and a second questionnaire to be completed during week 5 of the study. Each questionnaire takes about 10-20 minutes to complete.

**Watch videos**: You will watch 2 educational videos regarding air pollution exposure and its health effects and ways to reduce your exposure. Each video is between 3-5 minutes in length.

**Use air pollution sensor**: You will be provided with a Plume Labs Flow 2 air pollution sensor and a fanny pack free of charge that will be yours to keep even after the study ends. You will wear the Flow 2 personal air pollution sensor on a fanny pack from 9 a.m. to 9 p.m. PST over 5 weeks. You will be asked to send your air pollution measurements from the air pollution sensor each week for 5 weeks.

**Air quality text messages**: You will setup and receive EnviroFlash Air Quality Index (AQI) text alerts sent to your cell phone each day for 5 weeks. These alerts provide air pollution forecasts for the upcoming day.

You do not have to be in this study. You are free to say yes or no, or to drop out after joining. There is no penalty or loss of benefits for saying no or dropping out. Whatever you decide, your regular medical care will not change.

If you leave the study, your information cannot be removed from the study records.

# Protecting your Privacy as an Individual and the Confidentiality of Your Personal Information

Some organizations may need to look at your research records for quality assurance or data analysis. These include:

- Researchers involved with this study.
- The study sponsor and their agents.
- Fred Hutchinson Cancer Research Center.
- Institutional Review Boards (IRB), including the Fred Hutchinson Cancer Research Center IRB. An IRB is a group that reviews the study to protect your rights as a research participant.
- Office for Human Research Protections

We will assign a random number to your study record. The researchers conducting analyses with your information will not have access to your name or other personal information. They will know the random number only. Thus, the risk of someone connecting any study information with you as an individual is unlikely.

We will keep your records confidential. We will not use your personal information in any reports about this study such as journal articles or presentations at scientific meetings.

#### Other information.

After about 5 years, your personal information in the database will be destroyed.

If you have questions or complaints about this study, please call Dr. Trang VoPham at 206-667-2642. If you have questions about your rights as a research participant, call the Director of the Fred Hutch Institutional Review Office at 206-667-5900 or email irodirector@fredhutch.org.

The physical risks of this study are minimal. However, there is a very small risk inherent in any type of data collection that your confidentiality may be compromised. Any collected information will be stored in a secure location with restricted access. Any collected information will be kept separate from your name.

## Will I be paid to take part in this research study?

The entire study will be completed in 5 weeks and there are no costs for participating in this study. You will be given \$50 for completing each of the study tasks, totaling \$350.

## Do I have to participate in the whole study?

Each part of the study is completely voluntary. You may choose to join all, some, or none of the study activities. You may choose not to answer some questions.

#### Will you contact me in the future?

No.

## What will my information be used for?

Your information will only be used for the purposes of this study. Only authorized study staff will have access to your data. Data collected from this study will provide valuable information regarding how to best inform people about their air pollution exposure and potential health risks.

| Do you consent to be in | this study? | |
|---|---|---|
| ☐ Yes | | |
| $\square$ No | | |
| <ul><li>had the oppor</li><li>had the oppor</li><li>and</li></ul> | form (or had it read to you);<br>tunity to ask any questions you have<br>tunity to discuss the research with<br>sipate in this study. | |
| Participant: | | |
| Printed Name | Signature | Date |